CLINICAL TRIAL: NCT06816888
Title: Impact of Automatic Prompts in Echocardiographic Reports on Referral to Cardiology - A Randomized Control Study
Brief Title: Impact of Automatic Prompts in Echocardiographic Reports on Referral to Cardiology
Acronym: Echo Prompts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20240570-01H
Record Dates: First submitted 2025-01-29; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Mitral Regurgitation (MR); Moderate or Severe Aortic Stenosis (AS) (Mean Pressure Gradient ≥ 20 mm Hg or Aortic Valve Area ≤ 1.5 cm2)
Keywords: Echo prompts; valvular heart disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Lymphoma, Follicular; Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 3 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention arm 1 (Active Comparator): In this case, the prompt included will say "Your patient has been diagnosed with a moderate / severe valvular heart disease. Consider referral to a Cardiologist."
  Interventions: Other: Prompt 1
- Intervention arm 2 (Active Comparator): In this case, the prompt included will say "Your patient has been diagnosed with a moderate /severe valvular heart disease. Consider referral to the UOHI Center for Valvular Heart Disease".
  Interventions: Other: Prompt 2
- Control arm (Placebo Comparator): In this case no prompt will be added.
  Interventions: Other: No Prompt

INTERVENTIONS:
Other: No Prompt — Presence and type of message included in the prompt will be randomized
  Arms: Control arm
Other: Prompt 1 — Presence and type of message included in the prompt will be randomized
  Arms: Intervention arm 1
Other: Prompt 2 — Presence and type of message included in the prompt will be randomized
  Arms: Intervention arm 2

SUMMARY:
Echo Prompts study is a multi-center randomized controlled study to evaluate the impact of automatic prompts added to the conclusion of the echocardiographic reports of patient diagnosed with significant VHD 1) suggesting referral to a cardiologist or 2) suggesting referral to a cardiologist and offering the help of the University of Ottawa Heart Institute Center for Valvular Heart Diseases, compared to current standard of care (no prompts) on the rates and time to an evaluation by a cardiologist. We plan to involve a total of 300 patients in total. Primary endpoint will be the rate of referrals of patients having VHD to a cardiologist within 6 months after their TTE.

DETAILED DESCRIPTION:
Valvular heart disease (VHD) is next epidemic in the cardiovascular field, affecting millions of people worldwide and having a major impact on health care systems. With aging of the population, the incidence and prevalence of VHD will continue to increase.1-3 There is no medication that can prevent VHD progression. Appropriate management of patients with VHD relies on 3 pillars, early diagnosis, careful follow-up, and timely intervention. Regular follow-up by cardiologists and implementation of specialized VHD clinics have demonstrated a beneficial effect on patients' outcomes. 4Unfortunately, multiple studies have shown that patients with VHD remain undertreated and referred late in the course of the disease with inequality in access to care and treatment options. 5-12 Late presentation is associated with major penalties for patients who incur an increased risk of mortality and morbidity not restored even by a successful intervention. 13-17 In a community-based study collecting all consecutive patients diagnosed with moderate or severe mitral regurgitation (MR) based on echocardiography, only 15% were referred to surgery despite a clear (class I) indication for intervention. 18 These findings are even more remarkable as all patients were diagnosed with an echocardiogram performed at the Mayo Clinic, they had access to a world renown institution capable of achieving excellent surgical outcomes and there were no health care coverage issues. Potential reasons explaining the late referral and undertreatment of patients with VHD are insufficient physicians' knowledge regarding the management and timing of intervention, misbelief regarding the risk/benefit ratio of valvular interventions, incomplete understanding of the echocardiogram reports and limited access to cardiologists and more specifically to VHD specialists. 19, 20 We hypothesize that highlighting the importance of valvular echocardiographic findings to the ordering (non-cardiologist) physicians in an easy and comprehensive wording and offering access to cardiologists specialized in VHD will improve patients' referral rates to cardiologist and ultimately patients' outcomes. Implementation of prompts into clinical reports in various settings including VHD has been advocated but formal demonstration of its efficacy is lacking.

In this randomized controlled study, we will evaluate the impact of automatic prompts added to the conclusion of the echocardiographic reports of patient diagnosed with significant VHD 1) suggesting referral to a cardiologist or 2) suggesting referral to a cardiologist and offering the help of the University of Ottawa Heart Institute Center for Valvular Heart Diseases, compared to current standard of care (no prompts) on the rates and time to an evaluation by a cardiologist. This study will enable us to assess the impact of diagnostic prompts in isolation and associated to a facilitated access to VHD experts compared to our current practice.

This study is being conducted to see if addition of a prompt will increase the rate of patients seen by a cardiologist within 6 months after the TTE by 20% (absolute increase).

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. Patients diagnosed with moderate or severe aortic stenosis (AS) (mean pressure gradient ≥ 20 mm Hg or aortic valve area ≤ 1.5 cm2) or mitral regurgitation (MR) (based on integrative approach)
3. Patients referred by a non-cardiologist physician
4. Patients not currently followed by a cardiologist or who have seen a cardiologist within 24 months prior to the TTE

Exclusion Criteria:

1. Patients followed by a cardiologist or referred for a TTE by a Cardiologist
2. Less than moderate AS and MR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of referrals | 6 months
  The primary outcome measure of this study will be to compare the rates of patients seen by a cardiologist with 6 months between the 3 arms.

SECONDARY OUTCOMES:
Time interval | At 6 months after enrollment
  To compare the time interval in days between TTE and visit to a cardiologist between the 3 arms.

CONTACTS AND LOCATIONS:
Overall Officials: David Messika-Zeitoun, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided